CLINICAL TRIAL: NCT01295749
Title: Reduction of no Flow Time During Out of Hospital Cardiac Arrest by Using Laryngeal Tube for Airway Management by Nurses.
Brief Title: Effects of Laryngeal Tube Ventilation on no Flow Time During Out of Hospital Cardiac Arrest
Acronym: FLOWERS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DCIC - 1014
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; No Flow; Emergency; Nurse; laryngeal Tube
MeSH Terms: conditions — Heart Arrest; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ventilation by laryngeal tube (Active Comparator): ventilation by laryngeal tube and continuous chest compression
  Interventions: Device: laryngeal tube ventilation and continuous chest compression
- ventilation by bag valve mask (Sham Comparator): ventilation by bag valve mask and interrupted chest compression
  Interventions: Device: laryngeal tube ventilation and continuous chest compression

INTERVENTIONS:
Device: laryngeal tube ventilation and continuous chest compression — Comparison of no flow time between two strategies in out of hospital cardiac arrest
  Other Names: Laryngeal Tube LTD, VBM
  Arms: ventilation by laryngeal tube
Device: laryngeal tube ventilation and continuous chest compression — Comparison of no flow time between two strategies in out of hospital cardiac arrest
  Other Names: Laryngeal Tube LTD, VBM
  Arms: ventilation by bag valve mask

SUMMARY:
International recommendations stress on the importance of no flow time reduction in cardiac arrest management. In fact, no flow time is an independent factor of morbidity and mortality.

In France, cardiac arrests are treated by first responders (including emergency nurses) before the arrival of a mobile intensive care unit. Those first responders use bag-valve-mask for ventilation and therefore practice conventional CPR (30 chest compression / 2 ventilation rhythm). Laryngeal tube is a safe and efficient device in cardiac arrest ventilation. The purpose of our study is to compare the no flow time between two strategies of out of hospital cardiac arrest management by first responders: conventional CPR with bag-valve-mask ventilation vs. compression only CPR with Laryngeal Tube ventilation.

DETAILED DESCRIPTION:
Multicentric, prospective, controlled, randomized study with parallel groups in single blind.

Patients will be included in chronological periods to avoid selection biais (one month with the first medical device the next month with the other one). The determination of these periods will be centralized. The emergency vehicles will be supplied sufficiently with devices. This design has been chosen in order to answer to the emergency problem.

Patients will be included and ventilated by paramedical staff (first responders) before medical staff (Mobile Intensive Care Unit) intervention. Complete detailed information will be given to the patient or to the family and consent asked.

The comparison of no flow time between the two strategies in out of hospital cardiac arrest will be the following :

A : ventilation by bag valve mask and interrupted chest compression B : ventilation by laryngeal tube and continuous chest compression

ELIGIBILITY:
Inclusion Criteria:

* preliminary treatment of cardiac arrest by fire fighters (Basic Life support)
* more than 18 years
* patient affiliated to the social security system or equivalent

Exclusion Criteria:

* certain death
* patient deprived of freedom by judicial or administrative decision
* patient under legal protection
* Pregnancy, parturient or breast feeding
* facial trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
comparison of no flow time between two strategies | arrival of paramedical staff T0
  group A : ventilation by bag valve mask and interrupted chest compression group B : ventilation by laryngeal tube and continuous chest compression
  outcome measure : time of no flow during Resuscitation by trained paramedical staff in out of hospital cardiac arrest

SECONDARY OUTCOMES:
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  No flow proportion during resuscitation by paramedical staff after emergency training
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  no flow proportion on total resuscitation duration
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  number of failure installation after 2 tests
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  Time of device installation
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  chest expansion during insuflation (yes/no)
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  Mortality : spontaneous cardiac activity recovery, hospital admission, reanimation service or hospital exit date, survival at 28 days , CPC evaluation for patients alive
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  incident during ventilation :
  obstruction number of manipulations to optimize ventilation
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  ETCO2
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest at T0
  Number of external electric shocks
qualitative observation of laryngeal tube use for ventilation of patients in cardiac arrest | during cardiac arrest a T0
  degradation due to technical manipulations

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Danel, MD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - SDIS, Fontaine, Isere
  - Samu Smur, Grenoble, Isere

REFERENCES:
- [Background] Nolan JP, Deakin CD, Soar J, Bottiger BW, Smith G; European Resuscitation Council. European Resuscitation Council guidelines for resuscitation 2005. Section 4. Adult advanced life support. Resuscitation. 2005 Dec;67 Suppl 1:S39-86. doi: 10.1016/j.resuscitation.2005.10.009. No abstract available. PMID 16321716
- [Background] Eftestol T, Sunde K, Steen PA. Effects of interrupting precordial compressions on the calculated probability of defibrillation success during out-of-hospital cardiac arrest. Circulation. 2002 May 14;105(19):2270-3. doi: 10.1161/01.cir.0000016362.42586.fe. PMID 12010909
- [Background] Eftestol T, Wik L, Sunde K, Steen PA. Effects of cardiopulmonary resuscitation on predictors of ventricular fibrillation defibrillation success during out-of-hospital cardiac arrest. Circulation. 2004 Jul 6;110(1):10-5. doi: 10.1161/01.CIR.0000133323.15565.75. Epub 2004 Jun 21. PMID 15210599
- [Background] Adrie C, Cariou A, Mourvillier B, Laurent I, Dabbane H, Hantala F, Rhaoui A, Thuong M, Monchi M. Predicting survival with good neurological recovery at hospital admission after successful resuscitation of out-of-hospital cardiac arrest: the OHCA score. Eur Heart J. 2006 Dec;27(23):2840-5. doi: 10.1093/eurheartj/ehl335. Epub 2006 Nov 2. PMID 17082207
- [Background] Edelson DP, Abella BS, Kramer-Johansen J, Wik L, Myklebust H, Barry AM, Merchant RM, Hoek TL, Steen PA, Becker LB. Effects of compression depth and pre-shock pauses predict defibrillation failure during cardiac arrest. Resuscitation. 2006 Nov;71(2):137-45. doi: 10.1016/j.resuscitation.2006.04.008. Epub 2006 Sep 18. PMID 16982127
- [Background] Abella BS, Sandbo N, Vassilatos P, Alvarado JP, O'Hearn N, Wigder HN, Hoffman P, Tynus K, Vanden Hoek TL, Becker LB. Chest compression rates during cardiopulmonary resuscitation are suboptimal: a prospective study during in-hospital cardiac arrest. Circulation. 2005 Feb 1;111(4):428-34. doi: 10.1161/01.CIR.0000153811.84257.59. PMID 15687130
- [Background] Wiese CH, Bahr J, Bergmann A, Bergmann I, Bartels U, Graf BM. [Reduction in no flow time using a laryngeal tube: comparison to bag-mask ventilation]. Anaesthesist. 2008 Jun;57(6):589-96. doi: 10.1007/s00101-008-1358-2. German. PMID 18338138
- [Background] Odegaard S, Pillgram M, Berg NE, Olasveengen T, Kramer-Johansen J. Time used for ventilation in two-rescuer CPR with a bag-valve-mask device during out-of-hospital cardiac arrest. Resuscitation. 2008 Apr;77(1):57-62. doi: 10.1016/j.resuscitation.2007.11.005. PMID 18164533
- [Background] Wik L, Kramer-Johansen J, Myklebust H, Sorebo H, Svensson L, Fellows B, Steen PA. Quality of cardiopulmonary resuscitation during out-of-hospital cardiac arrest. JAMA. 2005 Jan 19;293(3):299-304. doi: 10.1001/jama.293.3.299. PMID 15657322
- [Background] Abella BS, Alvarado JP, Myklebust H, Edelson DP, Barry A, O'Hearn N, Vanden Hoek TL, Becker LB. Quality of cardiopulmonary resuscitation during in-hospital cardiac arrest. JAMA. 2005 Jan 19;293(3):305-10. doi: 10.1001/jama.293.3.305. PMID 15657323
- [Background] Valenzuela TD, Kern KB, Clark LL, Berg RA, Berg MD, Berg DD, Hilwig RW, Otto CW, Newburn D, Ewy GA. Interruptions of chest compressions during emergency medical systems resuscitation. Circulation. 2005 Aug 30;112(9):1259-65. doi: 10.1161/CIRCULATIONAHA.105.537282. Epub 2005 Aug 22. PMID 16116053
- [Background] Kern KB, Hilwig RW, Berg RA, Ewy GA. Efficacy of chest compression-only BLS CPR in the presence of an occluded airway. Resuscitation. 1998 Dec;39(3):179-88. doi: 10.1016/s0300-9572(98)00141-5. PMID 10078808
- [Background] Berg RA, Sanders AB, Kern KB, Hilwig RW, Heidenreich JW, Porter ME, Ewy GA. Adverse hemodynamic effects of interrupting chest compressions for rescue breathing during cardiopulmonary resuscitation for ventricular fibrillation cardiac arrest. Circulation. 2001 Nov 13;104(20):2465-70. doi: 10.1161/hc4501.098926. PMID 11705826
- [Background] Yu T, Weil MH, Tang W, Sun S, Klouche K, Povoas H, Bisera J. Adverse outcomes of interrupted precordial compression during automated defibrillation. Circulation. 2002 Jul 16;106(3):368-72. doi: 10.1161/01.cir.0000021429.22005.2e. PMID 12119255
- [Background] Bowman FP, Menegazzi JJ, Check BD, Duckett TM. Lower esophageal sphincter pressure during prolonged cardiac arrest and resuscitation. Ann Emerg Med. 1995 Aug;26(2):216-9. doi: 10.1016/s0196-0644(95)70154-0. PMID 7618786
- [Background] Gabrielli A, Wenzel V, Layon AJ, von Goedecke A, Verne NG, Idris AH. Lower esophageal sphincter pressure measurement during cardiac arrest in humans: potential implications for ventilation of the unprotected airway. Anesthesiology. 2005 Oct;103(4):897-9. doi: 10.1097/00000542-200510000-00031. No abstract available. PMID 16192785
- [Background] Wenzel V, Idris AH, Banner MJ, Kubilis PS, Williams JL Jr. Influence of tidal volume on the distribution of gas between the lungs and stomach in the nonintubated patient receiving positive-pressure ventilation. Crit Care Med. 1998 Feb;26(2):364-8. doi: 10.1097/00003246-199802000-00042. PMID 9468177
- [Background] Wenzel V, Idris AH, Banner MJ, Kubilis PS, Band R, Williams JL Jr, Lindner KH. Respiratory system compliance decreases after cardiopulmonary resuscitation and stomach inflation: impact of large and small tidal volumes on calculated peak airway pressure. Resuscitation. 1998 Aug;38(2):113-8. doi: 10.1016/s0300-9572(98)00095-1. PMID 9863573
- [Background] Lawes EG, Baskett PJ. Pulmonary aspiration during unsuccessful cardiopulmonary resuscitation. Intensive Care Med. 1987;13(6):379-82. doi: 10.1007/BF00257678. PMID 3668071
- [Background] Sayre MR, Sakles JC, Mistler AF, Evans JL, Kramer AT, Pancioli AM. Field trial of endotracheal intubation by basic EMTs. Ann Emerg Med. 1998 Feb;31(2):228-33. PMID 9472186
- [Background] Bradley JS, Billows GL, Olinger ML, Boha SP, Cordell WH, Nelson DR. Prehospital oral endotracheal intubation by rural basic emergency medical technicians. Ann Emerg Med. 1998 Jul;32(1):26-32. doi: 10.1016/s0196-0644(98)70095-2. PMID 9656945
- [Background] Katz SH, Falk JL. Misplaced endotracheal tubes by paramedics in an urban emergency medical services system. Ann Emerg Med. 2001 Jan;37(1):32-7. doi: 10.1067/mem.2001.112098. PMID 11145768
- [Background] Dorges V, Wenzel V, Schumann T, Neubert E, Ocker H, Gerlach K. Intubating laryngeal mask airway, laryngeal tube, 1100 ml self-inflating bag-alternatives for basic life support? Resuscitation. 2001 Nov;51(2):185-91. doi: 10.1016/s0300-9572(01)00423-3. PMID 11718975
- [Background] Ocker H, Wenzel V, Schmucker P, Steinfath M, Dorges V. A comparison of the laryngeal tube with the laryngeal mask airway during routine surgical procedures. Anesth Analg. 2002 Oct;95(4):1094-7, table of contents. doi: 10.1097/00000539-200210000-00057. PMID 12351302
- [Background] Bein B, Carstensen S, Gleim M, Claus L, Tonner PH, Steinfath M, Scholz J, Dorges V. A comparison of the proseal laryngeal mask airway, the laryngeal tube S and the oesophageal-tracheal combitube during routine surgical procedures. Eur J Anaesthesiol. 2005 May;22(5):341-6. doi: 10.1017/s026502150500058x. PMID 15918381
- [Background] Genzwuerker HV, Finteis T, Slabschi D, Groeschel J, Ellinger K. Assessment of the use of the laryngeal tube for cardiopulmonary resuscitation in a manikin. Resuscitation. 2001 Dec;51(3):291-6. doi: 10.1016/s0300-9572(01)00410-5. PMID 11738781
- [Background] Figueredo E, Martinez M, Pintanel T. A comparison of the ProSeal laryngeal mask and the laryngeal tube in spontaneously breathing anesthetized patients. Anesth Analg. 2003 Feb;96(2):600-5, table of contents. doi: 10.1097/00000539-200302000-00054. PMID 12538219
- [Background] Mihai R, Knottenbelt G, Cook TM. Evaluation of the revised laryngeal tube suction: the laryngeal tube suction II in 100 patients. Br J Anaesth. 2007 Nov;99(5):734-9. doi: 10.1093/bja/aem260. Epub 2007 Sep 14. PMID 17872934
- [Background] Genzwuerker HV, Dhonau S, Ellinger K. Use of the laryngeal tube for out-of-hospital resuscitation. Resuscitation. 2002 Feb;52(2):221-4. doi: 10.1016/s0300-9572(01)00472-5. PMID 11841891
- [Background] Kette F, Reffo I, Giordani G, Buzzi F, Borean V, Cimarosti R, Codiglia A, Hattinger C, Mongiat A, Tararan S. The use of laryngeal tube by nurses in out-of-hospital emergencies: preliminary experience. Resuscitation. 2005 Jul;66(1):21-5. doi: 10.1016/j.resuscitation.2004.12.023. PMID 15993725
- [Background] Dorges V, Ocker H, Wenzel V, Sauer C, Schmucker P. Emergency airway management by non-anaesthesia house officers--a comparison of three strategies. Emerg Med J. 2001 Mar;18(2):90-4. doi: 10.1136/emj.18.2.90. PMID 11300206
- [Background] Dorges V, Wenzel V, Neubert E, Schmucker P. Emergency airway management by intensive care unit nurses with the intubating laryngeal mask airway and the laryngeal tube. Crit Care. 2000;4(6):369-76. doi: 10.1186/cc720. Epub 2000 Oct 13. PMID 11123878
- [Background] Asai T, Hidaka I, Kawachi S. Efficacy of the laryngeal tube by inexperienced personnel. Resuscitation. 2002 Nov;55(2):171-5. doi: 10.1016/s0300-9572(02)00170-3. PMID 12413755
- [Background] Asai T, Kawachi S. Use of the laryngeal tube by paramedic staff. Anaesthesia. 2004 Apr;59(4):408-9. doi: 10.1111/j.1365-2044.2004.03721.x. No abstract available. PMID 15023121
- [Background] Kurola J, Harve H, Kettunen T, Laakso JP, Gorski J, Paakkonen H, Silfvast T. Airway management in cardiac arrest--comparison of the laryngeal tube, tracheal intubation and bag-valve mask ventilation in emergency medical training. Resuscitation. 2004 May;61(2):149-53. doi: 10.1016/j.resuscitation.2004.01.014. PMID 15135191
- [Background] Kurola JO, Turunen MJ, Laakso JP, Gorski JT, Paakkonen HJ, Silfvast TO. A comparison of the laryngeal tube and bag-valve mask ventilation by emergency medical technicians: a feasibility study in anesthetized patients. Anesth Analg. 2005 Nov;101(5):1477-1481. doi: 10.1213/01.ANE.0000182330.54814.70. PMID 16244014
- [Background] Wiese CH, Bartels U, Schultens A, Steffen T, Torney A, Bahr J, Graf BM. Influence of airway management strategy on "no-flow-time" during an "advanced life support course" for intensive care nurses - a single rescuer resuscitation manikin study. BMC Emerg Med. 2008 Apr 10;8:4. doi: 10.1186/1471-227X-8-4. PMID 18402652
- [Background] Gueugniaud PY, David JS, Chanzy E, Hubert H, Dubien PY, Mauriaucourt P, Braganca C, Billeres X, Clotteau-Lambert MP, Fuster P, Thiercelin D, Debaty G, Ricard-Hibon A, Roux P, Espesson C, Querellou E, Ducros L, Ecollan P, Halbout L, Savary D, Guillaumee F, Maupoint R, Capelle P, Bracq C, Dreyfus P, Nouguier P, Gache A, Meurisse C, Boulanger B, Lae C, Metzger J, Raphael V, Beruben A, Wenzel V, Guinhouya C, Vilhelm C, Marret E. Vasopressin and epinephrine vs. epinephrine alone in cardiopulmonary resuscitation. N Engl J Med. 2008 Jul 3;359(1):21-30. doi: 10.1056/NEJMoa0706873. PMID 18596271
- [Background] Gueugniaud PY, Mols P, Goldstein P, Pham E, Dubien PY, Deweerdt C, Vergnion M, Petit P, Carli P. A comparison of repeated high doses and repeated standard doses of epinephrine for cardiac arrest outside the hospital. European Epinephrine Study Group. N Engl J Med. 1998 Nov 26;339(22):1595-601. doi: 10.1056/NEJM199811263392204. PMID 9828247
- [Background] Asai T, Moriyama S, Nishita Y, Kawachi S. Use of the laryngeal tube during cardiopulmonary resuscitation by paramedical staff. Anaesthesia. 2003 Apr;58(4):393-4. doi: 10.1046/j.1365-2044.2003.03095_15.x. No abstract available. PMID 12648133
- [Background] Asai T, Shingu K. The laryngeal tube. Br J Anaesth. 2005 Dec;95(6):729-36. doi: 10.1093/bja/aei269. PMID 16286348
- [Background] Cummins RO, Chamberlain DA, Abramson NS, Allen M, Baskett P, Becker L, Bossaert L, Delooz H, Dick W, Eisenberg M, et al. Recommended guidelines for uniform reporting of data from out-of-hospital cardiac arrest: the Utstein Style. Task Force of the American Heart Association, the European Resuscitation Council, the Heart and Stroke Foundation of Canada, and the Australian Resuscitation Council. Ann Emerg Med. 1991 Aug;20(8):861-74. No abstract available. PMID 1854070
- [Background] Lemaire F, Bion J, Blanco J, Damas P, Druml C, Falke K, Kesecioglu J, Larsson A, Mancebo J, Matamis D, Pesenti A, Pimentel J, Ranieri M; ESICM Task Force on Legislation Affecting Clinical Research in the Critically Ill Patient. The European Union Directive on Clinical Research: present status of implementation in EU member states' legislations with regard to the incompetent patient. Intensive Care Med. 2005 Mar;31(3):476-9. doi: 10.1007/s00134-005-2574-8. Epub 2005 Feb 15. No abstract available. PMID 15711974
- See also: Nom d'utilisateur : FLOWERS99 mot de passe : FLOWERSTST — https://www.clininfohosting.com/specif/FLOWERS/